CLINICAL TRIAL: NCT03147989
Title: A Parallel-Group Comparison of Two Doses Of Multihance (0.10 mmol/Kg and 0.05 mmol/Kg) When Used For Magnetic Resonance Imaging (MRI) of The Central Nervous System (CNS)
Brief Title: Retrospective Study of MRI With MULTIHANCE at 0.10 and 0.05 mmol/Kg Dose in CNS Patients
Status: Completed | Type: Observational
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: MH-151
Record Dates: First submitted 2017-04-14; First posted 2017-05-10 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-02

CONDITIONS: Central Nervous System Diseases; Central Nervous System Neoplasms
Keywords: MultiHance; MRI; CNS; Gadobenate Dimeglumine
MeSH Terms: conditions — Central Nervous System Diseases; Central Nervous System Neoplasms | interventions — gadobenic acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1, 0.10 mmol/kg: For patients having received MULTIHANCE at a standard dose of 0.10 mmol/kg for their clinically indicated MRI examination.
  Interventions: Drug: MultiHance
- Group 2, 0.05 mmol/kg: For patients having received MULTIHANCE at a dose of 0.05 mmol/kg for their clinically indicated MRI examination.
  Interventions: Drug: MultiHance

INTERVENTIONS:
Drug: MultiHance — gadolinium contrast agent
  Other Names: Gadobenate Dimeglumine

SUMMARY:
This is a retrospective study to collect already existing data and images from patients ≥ 2 years of age who had MRI for CNS diseases with MultiHance administration at a standard 0.10 mmol/kg dose or the half dose of 0.05 mmol/kg. The MRI images of all included patients will be prospectively reviewed in a blinded read to compare the efficacy of the two doses.

DETAILED DESCRIPTION:
This study is retrospective in design in that the MR images and other patient data, such as demographic data, will be collected from existing data for the selected patients meeting the inclusion criteria defined in this protocol. The study will be a multicenter study comparing interindividually two groups, one group of patients having received MULTIHANCE at a standard dose of 0.10 mmol/kg and the other group a dose of 0.05 mmol/kg for their clinically indicated MRI examination.

In order to minimize selection bias, recruitment will start with the "Final Date" of this protocol and, working backward chronologically from all the MR examinations stored in the local site Picture Archiving and Communication Systems (PACS), every patient meeting the inclusion criteria will be recruited for the study until the total number of patients (160) in each group will be reached.

The images of all included patients will be prospectively reviewed in a blinded read.

ELIGIBILITY:
Inclusion Criteria:

* Was at least 2 years of age at the time of the MRI with MULTIHANCE injection at the dose of either 0.1 or 0.05 mmol/kg (±20% in volume administered).
* Has available demographic and safety data.
* Belongs to one of these 4 sub-groups:

  1. Had a documented known extra-axial lesion of the CNS and previously underwent MRI with a 1.5T magnet requiring an injection of 0.1 mmol/kg MULTIHANCE.
  2. Had a documented known extra-axial lesion of the CNS and previously underwent MRI with a 1.5T magnet requiring an injection of 0.05 mmol/kg MULTIHANCE.
  3. Had a documented known lesion of the CNS (including extra-axial) and previously underwent MRI with 3T magnet requiring an injection of 0.1 mmol/kg MULTIHANCE.
  4. Had a documented known lesion of the CNS (including extra-axial) and previously underwent MRI with 3T magnet requiring an injection of 0.05 mmol/kg MULTIHANCE.
* Have both pre- and post-dose T1 SE/FSE, and/or GRE, and T2 SE/FSE, and FLAIR MR Images (when available).
* Has one of the two documented doses of MULTIHANCE (either 0.05 or 0.1 mmol/kg) administered for their MRI exam and/or the volume (mL) and weight of the patient available to be used to calculate the exact dose (mmol/kg) of MULTIHANCE that was administered.

Exclusion Criteria:

* Any patient who does not fulfill all of the inclusion criteria;
* Any patient who has been previously entered into this study. Patients must be enrolled only once into the study. Working backward chronologically from date of the final Protocol, if a patient has already been enrolled and appears in the PACs System again due to an earlier MRI, this patient must be excluded from the study (i.e., only the first qualifying MRI working backward chronologically from the date of the final Protocol should be included into the study).

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients ≥ 2 years of age, having had a Multihance administration with either a dose of 0.10 mmol/kg or a dose of 0.05 mmol/kg for MRI of the CNS for a suspected or known extra-axial tumor at 1.5T, or suspected or known CNS disease at 3.0T.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Non-inferiority in border delineation of lesions | 1 Day
  To show non-inferiority of a 0.05 mmol/kg dose of MULTIHANCE as compared to 0.10 mmol/kg dose of MULTIHANCE, in patients undergoing contrast-enhanced MRI of the CNS in terms of lesion visualization based on pre-dose + post-dose: Border delineation of lesions
Non-inferiority in visualization of internal morphology of lesions | 1 Day
  To show non-inferiority of a 0.05 mmol/kg dose of MULTIHANCE as compared to 0.10 mmol/kg dose of MULTIHANCE, in patients undergoing contrast-enhanced MRI of the CNS in terms of lesion visualization based on pre-dose + post-dose: visualization of internal morphology of lesions
Non-inferiority in contrast enhancement of lesions | 1 Day
  To show non-inferiority of a 0.05 mmol/kg dose of MULTIHANCE as compared to 0.10 mmol/kg dose of MULTIHANCE, in patients undergoing contrast-enhanced MRI of the CNS in terms of lesion visualization based on pre-dose + post-dose: contrast enhancement of lesions

SECONDARY OUTCOMES:
Comparison of patient level change in border delineation of lesions | 1 Day
  To compare the efficacy of MULTIHANCE in MRI of the CNS in patients at a dose of 0.10 mmol/kg and 0.05 mmol/ kg in terms of patient level changes from pre-dose to pre + post-dose, with regard to border delineation of lesions.
Comparison of patient level change in visualization of internal morphology of lesions | 1 Day
  To compare the efficacy of MULTIHANCE in MRI of the CNS in patients at a dose of 0.10 mmol/kg and 0.05 mmol/kg in terms of patient level changes from pre-dose to pre + post-dose, with regard to visualization of internal morphology of lesions
Comparison of patient level change in contrast enhancement of lesions | 1 Day
  To compare the efficacy of MULTIHANCE in MRI of the CNS in patients at a dose of 0.10 mmol/kg and 0.05 mmol/kg in terms of patient level changes from pre-dose to pre + post-dose, with regard to contrast enhancement of lesions
Comparison of Lesion-to-brain ratio | 1 Day
  To compare the two doses of MultiHance in terms of predose to postdose by lesion changes for up to the 3 largest lesions in Lesion-to-brain ratio
Comparison of contrast-to-noise ratio | 1 Day
  To compare the two doses of MultiHance in terms of predose to postdose by lesion changes for up to the 3 largest lesions in Contrast-to-noise ratio

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Priovano, MD, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Sarasota Memorial Hospital, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No